CLINICAL TRIAL: NCT03579537
Title: Effects of Exercise on Physical Fitness Among Hemodialysis Patients With Chronic Kidney Disease - as Part of the Project to Implement Exercise During Hemodialysis Reference 15/10
Brief Title: Effects of Exercise on Physical Fitness Among Hemodialysis Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Universidad Europea de Madrid (Other); Fundación Renal Iñigo Alvarez De Toledo (Other)
Responsible Party: Principal Investigator, Marcela Gonzalez Gross, Full Professor for Sport Nutrition and Exercise Physiology, Universidad Politecnica de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Universidad Politécnica Madrid; MGGross (Other: Universidad Politécnica de Madrid); Margarita Pérez Ruiz (Other: Universidad Europea de Madrid)
Record Dates: First submitted 2018-05-18; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Hemolysis
Keywords: Hemodialysis; Klotho Protein; Excercise; Lifestyle condition
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Intervention Model Description: One group who perform 3 first month just with normal treatment of hemodialysis and the next 3 month exercise intervention. (6 months in total)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodyalisis patients (Experimental): group of patients in hemodialysis who performs the exercise program
  Interventions: Other: Intradyalisis without exercise programe; Other: Intradyalisis with exercise programe

INTERVENTIONS:
Other: Intradyalisis without exercise programe — patients on hemodialysis are evaluated with all the variables at first (T1) and without intervening in the treatment for 3 months they are evaluated again (T2).
Other: Intradyalisis with exercise programe — After 3 first month without intervention and also during the time of hemodialysis, the patients star the exercise programe, the first part of the session, an exercise was carried out for cardiovascular work (pedaling on ergometer) and muscle toning, with special attention to the muscular development of the lower limbs (exercises with elastic bands and / or weighted ankles). The session increased in duration and intensity as the physical action program progressed throughout the duration of the permitted period (3 months) and always attending to the individual needs of each subject. In addition, each of the participants will be given a series of recommendations of exercise practice to be carried out during non-hemodialysis days, in order to complement the work done during the sessions.3 month later the investigator evaluated all the variable again (T3)

SUMMARY:
Regular physical exercise was adapted to the situation of the patient with hemodialysis to help improve the quality of life of the patient

DETAILED DESCRIPTION:
It has been observed that programs that combine aerobic and resistance exercise can increase muscular strength and endurance, functional capacity and quality of life of patients in Hemodialysis. Aerobic exercise and muscular endurance during dialysis increase blood flow at the muscular level with an increase in capillary surface area, which dynamizes the flow of urea and toxins from the tissues to the vascular compartment, which could improve the effectiveness of dialysis In addition, moderate regular exercise can modulate the inflammatory response, which would be beneficial in patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Famel and male between 55 - 85 year old. in hemodyalisis treatment

Exclusion Criteria:

* Younger than 55 years and older than 85 years.
* Presenting myocardial infarction in the previous 6 weeks.
* Unstable angina to exercise or at rest.
* Recent cerebral vascular disease or with risk of recurrence.
* Musculoskeletal, respiratory (COPD with frequent decompensation).
* Hypertensive disorders, patients with peripheral vascular disease,
* Active liver disease.
* Osteoporosis diagnosed, in which the medical criterion is contraindicated physical exercise.
* Solution of problems of the following circumstances:
* Fraction of cardiac ejection <of 45%, Hb <of 10gr / dl.
* Problematic vascular access, both immature fistulas or with risk of extravasation and catheter dysfunctions of postural characteristics.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Biochemical values, Protein KLOTHO at 3 month and 6 month | baseline, 3 month and 6 month
  The measurement of Klotho in plasma (obtained from peripheral blood collected in tube with EDTA 3K anticoagulant) was performed by ELISA, with Well-wash 4 MK microplate washer (Thermo Electron Corporation) and Mutiskan EX microplate reader (Thermo Electron Corporation ), using the Human soluble α-Klotho Assay kit (Immuno-Biological Laboratories Co., Ltd, Japan). All samples were analyzed in duplicate following recommendations.

SECONDARY OUTCOMES:
Change from baseline in Physical performance sit and stand at 6 month | Baseline and 6 month
  patients' performance in the 10-repetition sit to stand (STS-10), The STS-10, an index of lower-extremity strength, measures the time (in seconds) required to perform 10 consecutive repetitions of sitting down and getting up from a chair. Participants began the test with their arm crossed on their chest and sitting with their back against the chair. They were instructed to perform the task "as fast as possible," starting and finishing at the sitting position. Time was measured with a stopwatch (ONstart 100, Geonaute, France) to the nearest 0.1 second.
Change from baseline in Physical performance 6MWT at 6 month | Baseline and 6 month
  The 6MWT was used as a marker of endurance capacity. It was performed on a 17-meter corridor with marks on every meter, and time was measured with a chronometer. (ONstart 100, Geonaute, France). Participants were asked to cover the longest distance possible during six minutes by walking (not running) continuously and turning around at the final mark. No verbal encouragement was given during the test; however, feedback regarding the remaining time was available. Participants were allowed to rest during the test, and to use any ambulation aid that they used during daily life.
Change from baseline in Physical performance handgrip force at 6 month | Baseline and 6 month
  Maximal isometric handgrip force has been suggested as a useful tool for the continuous assessment of muscle mass and function in dialysis patients. It was measured in both hands using a manual dynamometer (T.K.K.5401, Takei Scientific Instruments, Japan) while participants were in a standing position, with the arm extended and parallel to the body, and without moving the wrist. They performed two maximal repetitions with each hand interspersed with one-minute rests, and the mean of all four trials was analyzed.
Change from baseline in Mental and health status (Beck Depression Inventory) at 6 month | Baseline and 6 month
  Changes in depression symptoms were assessed using the Beck Depression Inventory (BDI). In this self-reported questionnaire 21 items are rated on a four-point severity scale and summed to give a total score, being a higher score suggestive of more severe depression. The BDI has proven a valid depression screening tool in dialysis patients, being one of the most commonly used questionnaires to assess this condition in this patient population. The Scale of this questionaire is: No depression (0 - 13 points); Low depression (14 - 19 points); moderate depression (20 - 28 points); several depression (≥29 points)
Change from baseline in Mental and health status (Health-related QoL <HRQoL> ) at 6 month | Baseline and 6 month
  Health-related QoL (HRQoL) was assessed using the Short-Form 12 (SF-12) health survey, a short version of the SF-36. A physical (PCS) and a mental component score (MCS) are calculated from this self-reported questionnaire. SF-12 has proven reliable and valid in dialysis patients, being associated with short-term and long-term mortality in this population. The questionnaire is divided into three dimensions which have the following scales: EQ-EVA (visual analog scale) scores from 0 to 100 where 0 is the worst health state imaginable and 100 the best state, EQ-Descriptive. Better state of health self-perceived (11111) and worse (33333) depending on the answers given in each one of the sections of the questionnaire and EQ-Index. Better health status: values of 1 or close to 1 and the states closest to death.
Change from baseline in Mental and health status (level of anxiety) at 6 month | Baseline and 6 month
  the State-Trait Anxiety Inventory (STAI), The score range ranges from 0 to 60 points, so that high scores reflect greater anxiety. The scores obtained are transformed into decatypes (10 decatypes).
Hemogram and Biochemical values , (hemoglobin, hematocrit and mean corpuscular volume ) | Baseline
  Red blood cells, hemoglobin, hematocrit and mean corpuscular volume were determined from whole blood anticoagulated with EDTA in a Sysmex XI-1000i hematological analyzer. with normal values for hemoglobin 14± 2 (g/dL) for women and of 16± 2 (g/dL) for men, for hematocrit 42± 5 % for women and of 47± 6 % for men and for corpuscular volumen 90 ± 7 (fL) for women and for men.
Hemogram and Biochemical values (Iron, albumin, calcium and phosporus) | Baseline
  Iron, albumin, calcium and phosphorus were made by spectrophotometry from serum in a Cobas Integra 400 device. , considered as normal values Total calcium mg/100 mL 8,5-10,5; Phosphorus mg/100 mL 2,2-4,4; albumin g/100 mL 3-5 and for Iron 60 a 170 mcg/dL
Hemogram and Biochemical values (Transferrin) | Baseline
  Transferrin was obtained in a Cobas Integra 400 device by immunoturbidimetry technique from serum, considered as normal values for men and women 200-400 mg/dL (23-45 mmol/L).
Hemogram and Biochemical values (Ferritin and PTH) | Baseline
  Ferritin and PTH were determined from serum by chemiluminescence technique using an Elecsys 2010 equipment. with normal values for ferritin 12-300 ng/mL for men and 12-200 ng/mL for women and for PTH 8 - 51 pg/mL (8 - 51 ng/L) for men and women.
Hemogram and Biochemical values (The ions (Na +, K + and Cl-)) | Baseline
  The ions (Na +, K + and Cl-) were determined in serum using a Cobas Integra 400 device by means of a selective electrode module.
Hemogram and Biochemical values (The transferrin saturation index (IST)) | Baseline
  The transferrin saturation index (IST) was obtained through the following formula: IST (%) = (serum iron concentration (M)) / (2 x transferrin concentration (M)) * 100. considered as normal values for men and women 20 - 50%
Change in Body Composition, Body mass index (BMI) | Baseline, 3 months and 6 ,months
  The age in years; height in centimeters (tallimeter Ano Sayol SL, Barcelona, Spain); weight in kilograms (Inbody 720, Microcaya) and we can derive from this data the variable of Body Mass Index (BMI) calculated as weight (kg)/height (m2).
Change in Body Composition, Body Fat Index | Baseline, 3 months and 6 ,months
  For determinate this variable of the body composition will be use a Bioelectrical impedance machine Inbody 720, Microcaya. The datas of Total Body Fat Index shown in percentage and kilograms.
Change in Body Composition, Fat Mass by body segment | Baseline, 3 months and 6 ,months
  For determinate this variable of the body composition will be use a Bioelectrical impedance machine Inbody 720, Microcaya. The datas of Fat Mass shown in kilograms. This is divided in upper limb and lower limb on both side (left and right) and Trunk Fat Mass.
Change in Body Composition, Total Muscle Mass | Baseline, 3 months and 6 ,months
  For determinate this variable of the body composition will be use a Bioelectrical impedance machine Inbody 720, Microcaya. The datas of Total Muscle Mass shown in kilograms. This is divided in upper limb and lower limb on both side (left and right) and Trunk Muscle Mass.
Sociocultural aspects | Baseline
  It is assumed that they are linked to the center where the study will be conducted. However, the EXERNET questionnaire will be included and it does not have cut points since it collects general and descriptive data of the subject.

IPD SHARING:
Plan to Share IPD: No